CLINICAL TRIAL: NCT00436839
Title: An Multicenter, Randomized Study of Comparison of Docetaxel Plus Prednisone With Mitoxantrone Plus Prednisone in the Patients With Hormone-refractory (Androgen-independent) Metastatic Prostate Cancer
Brief Title: Taxotere Prostate Cancer New Indication Registration Trial in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_01833
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Mitoxantrone; Prednisone

ARMS (2):
- 1 (Experimental): Docetaxel 75mg/m² intravenously (day 1) every 21 days, plus prednisone 10mg orally given daily, minimal for 6 cycles and up to 10 cycle
  Interventions: Drug: Docetaxel; Drug: Prednisone
- 2 (Active Comparator): Mitoxantrone 12mg/m² intravenously every 21 days, plus prednisone 10mg orally given daily, minimal for 6 cycles and up to 10 cycle
  Interventions: Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — 75mg/m² intravenously (day 1) every 21 days
  Arms: 1
Drug: Mitoxantrone — 12mg/m² intravenously every 21 days
  Arms: 2
Drug: Prednisone — 10mg orally given daily

SUMMARY:
To compare overall survival after receiving mitoxantrone and prednisone or docetaxel and prednisone in subjects with hormone-refractory metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven prostate adenocarcinoma
* Androgen independent prostate Cancer S/P orchiectomy and/or LHRH agonist Testosterone < 50 ng/dl (ie 1.735 nmol/l)
* Documented progressive disease
* Patients should have achieved stable analgesia for 7 days
* Karnofsky Performance Status ≥ 70
* No prior treatment with cytotoxic agent (except estramustine)
* Normal cardiac function must be confirmed by Left ventricular ejection fraction
* Adequate organ function:

  1. Hematology:

     * Neutrophils > 1.5 x 10^9/L
     * Hemoglobin > 10 g/dl. Erythropoietin use is allowed, but red blood cell transfusion to upgrade the hemoglobin level is not allowed
     * Platelets > 100 x 10^9/L
  2. Hepatic function:

     * Total bilirubin < the upper-normal limit of the institution.
     * Alanine aminotransferase and Aspartate transaminase < 1.5 times the upper-normal limit of the institution.
  3. Renal function:

     * Creatinine < 1.5 times the upper normal limit (ie National Cancer Institution grade < 1)
* No brain or leptomeningeal metastases

Exclusion Criteria:

* Prior radiotherapy to >25% of bone marrow (whole pelvic irradiation is not allowed)
* prior cytotoxic chemotherapy, except monotherapy with estramustine
* prior isotope therapy
* history of another cancer within the preceding five year
* symptomatic peripheral neuropathy grade ≥ 2
* other serious illness or medical condition:

  1. Congestive heart failure even if controlled. Previous history of myocardial infarction or angina pectoris within 1 year from study entry, uncontrolled hypertension or uncontrolled arrhythmias.
  2. Active uncontrolled infection
  3. Peptic ulcer, unstable diabetes mellitus or other contraindications for the use of corticosteroids.
  4. Auto-immune disease (lupus, sclerodermia, rheumatoid polyarthritis)
* treatment with any other anti-cancer therapy
* treatment with bisphosphonates

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy: Overall survival | From beginning to end of the study
Objective response rate of patients with measurable disease by Response Evaluation Criteria in Solid tumours | From beginning to end of study
Prostatic Specific Antigen response | From the beginning to the end of study
Pain response (McGill-Melzack Scale) | From beginning to end of study
Time to progression | From beginning to end of study
Adverse event | From beginning to end of study
Quality Of Life: Functional assessment of chronic illness therapy-prostate questionnaire will be used | From beginning to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jing Fu, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

REFERENCES:
- [Derived] Zhou T, Zeng SX, Ye DW, Wei Q, Zhang X, Huang YR, Ye ZQ, Yang Y, Zhang W, Tian Y, Zhou FJ, Jie J, Chen SP, Sun Y, Xie LP, Yao X, Na YQ, Sun YH. A multicenter, randomized clinical trial comparing the three-weekly docetaxel regimen plus prednisone versus mitoxantone plus prednisone for Chinese patients with metastatic castration refractory prostate cancer. PLoS One. 2015 Jan 27;10(1):e0117002. doi: 10.1371/journal.pone.0117002. eCollection 2015. PMID 25625938